CLINICAL TRIAL: NCT04845542
Title: Testing Efficacy of an Intervention to Promote Resilience in Stroke Survivor-carepartner Dyads (ReStoreD)
Brief Title: Promoting Resilience in Stroke Survivor-carepartner Dyads (ReStoreD)
Acronym: ReStoreD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Alexandra Terrill, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01HD105718-01 (NIH)
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Depression, Anxiety; Coping Skills; Couples
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized waitlist control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReStoreD (Experimental): 8-week intervention that is remotely delivered, consisting of psychoeducation and positive psychology activities. Participants complete two activities individually and two together each week.
  Interventions: Behavioral: ReStoreD
- Waitlist-control (No Intervention): Participants will be waitlisted for 8 weeks.

INTERVENTIONS:
Behavioral: ReStoreD — ReStoreD is a remotely-administered behavioral intervention in which couples coping with stroke learn and practice goal-setting, communication strategies, and positive psychology activities, such as expressing gratitude, finding meaning, and fostering connections. Participants are provided with 8 weekly modules, each featuring two components: 1) psychoeducational materials, such as an informational video and resources/links about a general topic related to resilience, coping, and/or overall well-being of the individual and couple, and 2) examples of positive psychology activities that relate to the week's theme or topic. Participants are asked to complete at least two positive psychology activities alone and two together each week.
  Arms: ReStoreD

SUMMARY:
Affecting nearly 800,000 people in the US every year, stroke is a leading cause of long-term disability, and has serious consequences for stroke survivors and their carepartners. Our project uses a scientifically rigorous efficacy study to evaluate a remotely delivered 8-week dyadic (couples-based) positive psychology intervention to reduce emotional distress in stroke survivors and their carepartners. If successful, couples may be better emotionally equipped to cope with the sequelae of stroke, and have better rehabilitation outcomes and quality of life.

DETAILED DESCRIPTION:
The impact of stroke is shared between the stroke survivor and their spousal/partner caregiver (carepartner). An estimated 30-50% of stroke survivors and carepartners experience depressive or anxiety symptoms that negatively affect rehabilitation outcomes and quality of life. Yet, interventions to support couples post-stroke are largely insufficient or inaccessible. To address this need, we developed a novel remotely-delivered dyadic intervention to promote Resilience in Stroke survivor-carepartner Dyads (ReStoreD), in which couples learn and practice goal-setting, communication strategies, and positive psychology activities like expressing gratitude, finding meaning, and fostering connections. Preliminary pilot study results were promising, showing reduced depressive symptoms and increased resilience in participants. The purpose of the current study is to conduct a Stage II efficacy trial of the 8-week ReStoreD intervention with a sample of 200 dyads (n=400) consisting of one individual who has sustained an ischemic or hemorrhagic stroke between 3 months and 3 years prior to enrollment and a cohabitating carepartner. Using a fully-powered, randomized waitlist-control design, we will determine efficacy of ReStoreD to reduce emotional distress in both dyad members (Aim 1). We will also examine effects of ReStoreD on secondary outcomes (resilience, relationship quality, stress-related stroke, meaningful activity engagement) as potential mediators (Aim 2), and explore moderators to determine whether certain subgroups respond better to the intervention (Aim 3). All participants will complete standardized, validated assessments at baseline, 8 weeks, 16 weeks, and 6-month follow up. All aspects of the study, including intervention activities and assessments, are conducted remotely, online.

This is the first rigorously designed efficacy trial to test a positive psychology intervention for stroke survivors and their carepartners. When the aims of this study are realized, we will 1) have a remotely-delivered, dyadic intervention to support couples post-stroke; 2) have a better understanding of the mechanisms involved in the intervention's effect on emotional distress, and can use this information to inform future interventions; and 3) be able to identify a more specific target population for whom the intervention works best. Ultimately, if found efficacious, this intervention will offer sustainable and accessible support for couples who are coping with stroke to improve rehabilitation outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling cohabitating couple where one partner has a had an ischemic or hemorrhagic stroke
* The stroke must have occurred between 3 months and 3 years prior to enrollment
* The adult couple must have been living together since before the stroke and for at least 6 months prior to enrollment
* One or both partners must report some anxiety and/or depressive symptoms
* Participants must be able to read, understand, and follow instructions, and be able to provide their own consent

Exclusion Criteria:

• Either dyad partner has significant aphasia (difficulties with speech), visual, psychiatric, and/or significant cognitive impairment that would limit their ability to participate in the intervention in a meaningful way

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Emotional Distress, Anxiety and Depression Scale-Short Form | Baseline
  8-item self-report measure of depression (4 items) and anxiety (4 items); higher scores indicate more emotional distress
PROMIS Emotional Distress, Anxiety and Depression Scale-Short Form | 8 weeks
  8-item self-report measure of depression (4 items) and anxiety (4 items); higher scores indicate more emotional distress
PROMIS Emotional Distress, Anxiety and Depression Scale-Short Form | 16 weeks
  8-item self-report measure of depression (4 items) and anxiety (4 items); higher scores indicate more emotional distress
PROMIS Emotional Distress, Anxiety and Depression Scale-Short Form | 6 months
  8-item self-report measure of depression (4 items) and anxiety (4 items); higher scores indicate more emotional distress

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | baseline
  10-item self-report measure of resilience; higher scores indicate greater resilience
Connor-Davidson Resilience Scale (CD-RISC) | 8 weeks
  10-item self-report measure of resilience; higher scores indicate greater resilience
Connor-Davidson Resilience Scale (CD-RISC) | 16 weeks
  10-item self-report measure of resilience; higher scores indicate greater resilience
Connor-Davidson Resilience Scale (CD-RISC) | 6 months
  10-item self-report measure of resilience; higher scores indicate greater resilience
Dyadic Coping Inventory (DCI)-short | baseline
  11-item self-report measure of how well the couple copes with stress; higher scores indicate better coping
Dyadic Coping Inventory (DCI)-short | 8 weeks
  11-item self-report measure of how well the couple copes with stress; higher scores indicate better coping
Dyadic Coping Inventory (DCI)-short | 16 weeks
  11-item self-report measure of how well the couple copes with stress; higher scores indicate better coping
Dyadic Coping Inventory (DCI)-short | 6 months
  11-item self-report measure of how well the couple copes with stress; higher scores indicate better coping
Dyadic Relationship Scale | baseline
  Self report measure that assesses care-recipient-caregiver relationship and includes 2 subscales: Dyadic Strain (5 items; higher scores mean more strain) and Positive Dyadic Interactions (6 items; higher scores mean more positive interactions)
Dyadic Relationship Scale | 8 weeks
  Self report measure that assesses care-recipient-caregiver relationship and includes 2 subscales: Dyadic Strain (5 items; higher scores mean more strain) and Positive Dyadic Interactions (6 items; higher scores mean more positive interactions)
Dyadic Relationship Scale | 16 weeks
  Self report measure that assesses care-recipient-caregiver relationship and includes 2 subscales: Dyadic Strain (5 items; higher scores mean more strain) and Positive Dyadic Interactions (6 items; higher scores mean more positive interactions)
Dyadic Relationship Scale | 6 months
  Self report measure that assesses care-recipient-caregiver relationship and includes 2 subscales: Dyadic Strain (5 items; higher scores mean more strain) and Positive Dyadic Interactions (6 items; higher scores mean more positive interactions)
PROMIS-Psychosocial Illness Impact Scale-short form | baseline
  8-item self report measure on stroke-related stress (completed by person with stroke only); higher scores indicate greater negative impact/more stress.
PROMIS-Psychosocial Illness Impact Scale-short form | 8 weeks
  8-item self report measure on stroke-related stress (completed by person with stroke only); higher scores indicate greater negative impact/more stress.
PROMIS-Psychosocial Illness Impact Scale-short form | 16 weeks
  8-item self report measure on stroke-related stress (completed by person with stroke only); higher scores indicate greater negative impact/more stress.
PROMIS-Psychosocial Illness Impact Scale-short form | 6-months
  8-item self report measure on stroke-related stress (completed by person with stroke only); higher scores indicate greater negative impact/more stress.
Zarit Burden Inventory-Short | baseline
  12 item self-report measure on caregiving related stress/burden (completed by partner only); higher scores indicate more burden
Zarit Burden Inventory-Short | 8 weeks
  12 item self-report measure on caregiving related stress/burden (completed by partner only); higher scores indicate more burden
Zarit Burden Inventory-Short | 16 weeks
  12 item self-report measure on caregiving related stress/burden (completed by partner only); higher scores indicate more burden
Zarit Burden Inventory-Short | 6 months
  12 item self-report measure on caregiving related stress/burden (completed by partner only); higher scores indicate more burden
Meaningful Activity Participation Assessment (MAPA) | baseline
  28 activity items are rated on frequency of engaging in these activities (higher score means more frequent) and how meaningful they are to the person (higher score means more meaningful)
Meaningful Activity Participation Assessment (MAPA) | 8 weeks
  28 activity items are rated on frequency of engaging in these activities (higher score means more frequent) and how meaningful they are to the person (higher score means more meaningful)
Meaningful Activity Participation Assessment (MAPA) | 16 weeks
  28 activity items are rated on frequency of engaging in these activities (higher score means more frequent) and how meaningful they are to the person (higher score means more meaningful)
Meaningful Activity Participation Assessment (MAPA) | 6 months
  28 activity items are rated on frequency of engaging in these activities (higher score means more frequent) and how meaningful they are to the person (higher score means more meaningful)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Terrill, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No